CLINICAL TRIAL: NCT05194423
Title: THE TRAVEL II TRIAL: Transcatheter Right Atrial-ventricular Valve rEplacement With LuX-Valve Via Jugular Vein
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Fu Wai Hospital, Beijing, China (Other); Beijing Anzhen Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); Xijing Hospital (Other); Guangdong Provincial People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhiyun Xu, Chair of Department of Cardiovascular Surgery, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAVEL II
Record Dates: First submitted 2021-12-28; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Tricuspid Valve Regurgitation
Keywords: Tricuspid valve regurgitation; Transcatheter tricuspid valve replacement; LuX-Valve
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center single-arm trial in eight centers in China. A minimum of 150 subjects will be enrolled in this study and followed-up at discharge (≤ 10 days post operation), 30 days, 6 months, 1, 2, 3, 4, 5 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tricuspid Valve Replacement System via jugular vein (Experimental): Subjects who received transcatheter tricuspid valve replacement with LuX-Valve and delivery system via jugular vein will be included in this arm.
  Interventions: Device: Tricuspid Valve Replacement System via jugular vein

INTERVENTIONS:
Device: Tricuspid Valve Replacement System via jugular vein — To eliminate the tricuspid regurgitation through orthotopically replacing tricuspid valve with LuX-Valve system via jugular vein.

SUMMARY:
The trial aims to evaluate the safety and effectiveness of LuX-Valve transcatheter tricuspid valve and delivery system via jugular vein which are intended to use in symptomatic patients with severe tricuspid regurgitation and high surgical risk.

DETAILED DESCRIPTION:
The TRAVEL II study is a prospective multi-center single-arm trial for transcatheter tricuspid valve replacement with LuX-Valve via jugular vein. A series of physical, imaging and laboratory exams will be performed to determine whether a subject has severe tricuspid regurgitation with high surgical risk. Subjects who meet the criteria will then receive LuX-Valve implantation via jugular vein if an informed consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years at time of consent.
2. Subjects or subject's legal representative has been informed of the nature of the study and provided written informed consent.
3. The site heart team confirmed the subject is at high risk for tricuspid valve surgery (euroSCORE II ≥ 7.0%) and the subject will get benefit from the intervention.
4. Subjects must guarantee they won't participate in any other clinical trial for a period of one year after the intervention.
5. Subjects are with New York Heart Association (NYHA) Functional Class III or IV.
6. Subjects are with normal left heart function (EF ≥ 50%).
7. No indications for left-sided or pulmonary valve intervention.
8. Subjects must have severe or greater tricuspid regurgitation ( the vena contracta (VC) width ≥ 7 mm or the effective regurgitant orifice area (EROA) ≥ 40 mm2), which confirmed by the Echocardiography Core Lab (ECL) via transthoracic echocardiogram (TTE).

Exclusion Criteria:

1. Subjects with pulmonary hypertension (systolic pressure ≥ 55mmHg determined by right heart catheterization).
2. Subjects with previous transcatheter or surgical tricuspid valve procedure.
3. Subjects with tricuspid stenosis or other anatomy disorders that unsuitable for the procedure.
4. Subjects with depressed right heart function (tricuspid annular plane systolic excursion (TAPSE) < 10mm or right ventricle fractional area change (FAC) < 20%).
5. Subjects with aortic stenosis (mean ΔP≥ 40mmHg or aortic valve area ≤ 1 cm2), aortic regurgitation (≥ 3+), mitral stenosis (mitral valve area ≤1.5 cm2) or mitral regurgitation (≥ 3+).
6. Subjects with active endocarditis or other infectious diseases.
7. Subjects with untreated severe coronary artery disease.
8. Subjects with percutaneous coronary intervention, cerebrovascular accident or surgical intervention within 3 months of the date of the procedure.
9. Subjects with coagulation disorders.
10. Subjects with known allergy, hypersensitivity or contraindication to the material or drugs used in the procedure.
11. Subjects with cognitive disorders that can not cooperate the study or follow-up.
12. Subjects with less than 12 months life expectancy because of non-cardiac conditions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Death | 1 year
  All-cause Death
Tricuspid Regurgitation Reduction | 1 year
  Tricuspid regurgitation measured with echocardiography in core lab reduces at least 2 grades.

SECONDARY OUTCOMES:
Device or Procedure-Related Adverse Events | 1 year
  Device related mortality, device malposition, right ventricular outflow tract obstruction, conduction system disturbances, new onset shunt across ventricular septum, coronary artery injury, valve failure, convert to open surgery, reintervention, embolization.
Device or Procedure-Related Adverse Events | 2 year
  Device related mortality, device malposition, right ventricular outflow tract obstruction, conduction system disturbances, new onset shunt across ventricular septum, coronary artery injury, valve failure, convert to open surgery, reintervention, embolization.
Device or Procedure-Related Adverse Events | 3 year
  Device related mortality, device malposition, right ventricular outflow tract obstruction, conduction system disturbances, new onset shunt across ventricular septum, coronary artery injury, valve failure, convert to open surgery, reintervention, embolization.
Device or Procedure-Related Adverse Events | 4 year
  Device related mortality, device malposition, right ventricular outflow tract obstruction, conduction system disturbances, new onset shunt across ventricular septum, coronary artery injury, valve failure, convert to open surgery, reintervention, embolization.
Device or Procedure-Related Adverse Events | 5 year
  Device related mortality, device malposition, right ventricular outflow tract obstruction, conduction system disturbances, new onset shunt across ventricular septum, coronary artery injury, valve failure, convert to open surgery, reintervention, embolization.
Major Adverse Event (MAE) | 1 year
  MAE includes death, myocardial infarction, stroke, reoperation for bleeding, renal failure, pulmonary embolism, gastrointestinal hemorrhage, rehospitalization.
Major Adverse Event (MAE) | 2 year
  MAE includes death, myocardial infarction, stroke, reoperation for bleeding, renal failure, pulmonary embolism, gastrointestinal hemorrhage, rehospitalization.
Major Adverse Event (MAE) | 3 year
  MAE includes death, myocardial infarction, stroke, reoperation for bleeding, renal failure, pulmonary embolism, gastrointestinal hemorrhage, rehospitalization.
Major Adverse Event (MAE) | 4 year
  MAE includes death, myocardial infarction, stroke, reoperation for bleeding, renal failure, pulmonary embolism, gastrointestinal hemorrhage, rehospitalization.
Major Adverse Event (MAE) | 5 year
  MAE includes death, myocardial infarction, stroke, reoperation for bleeding, renal failure, pulmonary embolism, gastrointestinal hemorrhage, rehospitalization.
Functional Change in New York Heart Association (NYHA) Classification | 1 year
  Subjects' heart function is ranged from NYHA I to IV based on how much a patient is limited during physical activity. NYHA I means no limited on physical activity while NYHA IV means unable to take any physical activity.
Change in Quality of Life (QOL) is evaluated with Kansas City Cardiomyopathy (KCCQ) | 1 year
  KCCQ score ranges from 0 to 100, which 0 reflects the worst health status and 100 reflects the best health status.
Change in Quality of Life (QOL) is evaluated with Six Minute Walk Test (6MWT) | 1 year
  6MWT distance is recorded and compared with baseline during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyun Xu, MD, Principal Investigator — Changhai Hospital; Fanglin Lu, MD, Study Director — Changhai Hospital; Junbo Ge, MD, Principal Investigator — Shanghai Zhongshan Hospital; Shengshou Hu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (9):
- China (9):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Fu Wai Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xijing Hospital, Xi'an, Shaanxi
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No